CLINICAL TRIAL: NCT07130838
Title: Effects of Application-Based Mindfulness and Eating Awareness Training on Disordered Eating in Youth With Obesity: The MB-EAT Study
Brief Title: The MB-EAT Smart Teen Study
Acronym: MB-EAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gary Goldfield (Other)
Responsible Party: Sponsor-Investigator, Gary Goldfield, Senior Scientist, Children's Hospital of Eastern Ontario
Organization: Children's Hospital of Eastern Ontario (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OBIMBEAT25
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Feasibility Studies

STUDY DESIGN:
Intervention Model Description: Phase 1: Single arm intervention Phase 2: Parallel arm intervention
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1: Feasibility study (Experimental): Patients in the feasibility study will receive a modified, shortened version of the MB-EAT program through AmDTx-Epiq within the AmDTx app.
  Interventions: Behavioral: Feasibility study
- Phase 2: Control group Arm (Active Comparator): Patients allocated to the control group will receive audio-recorded psychoeducation consisting of standard diet/exercise information through the same AmDTx-Epiq in the AmDTx app.
  Interventions: Behavioral: Psychoeducation
- Phasee 2: Intervention group (Experimental): Patients allocated to the intervation arm will receive the manualized and audio-recorded MB-EAT program which will be delivered through modules in the form of a "journey" in the AmDTx app.
  Interventions: Behavioral: MB-EAT program

INTERVENTIONS:
Behavioral: MB-EAT program — Phase 2 will include 12 modules, delivered across 12 weeks. The program will contain seated and guided mindfulness practices designed to cultivate better awareness of hunger cues, sensory-specific satiety, as well as external and emotional food-related triggers through body scans, taste satiety and mindful eating practices, self-compassion meditations, and diaphragmatic breathing. The intervention will also include mindful movements. Each session will be focused on a specific theme related to promoting healthy eating behaviours and emotional regulation. Each module will be unlocked as the participant progresses through the program. AmDTx-Epiq also incorporates goal setting, daily feedback, prompts for change, and positive reinforcement in the form of an encouraging text messages from the study coach.
  Arms: Phasee 2: Intervention group
Behavioral: Feasibility study — Phase 1 will include 4 modules, delivered across 4 weeks. All participants will receive a modified, shortened version of the MB-EAT program through AmDTx-Epiq within the AmDTx app. Participants will also complete the "Keep in Balance" questionnaire every week on the app, a questionnaire which assesses weekly physically activity and eating habits, as well as associated thoughts and feelings to these. Participants will receive regular "check-ins" twice per week from a coach (unblinded study coordinator) via text designed to promote engagement and answer questions participants may have during the 4-week intervention period.
  Arms: Phase 1: Feasibility study
Behavioral: Psychoeducation — Patients in the control group will receive audio-recorded psychoeducation in the form of standard diet/exercise information. The comparator is publicly available psychoeducational information available on nutrition, physical activity, and weight management through best practice guidelines, clinical guidelines, and public health guidelines. These comparators were chosen as they are easily accessible standard of care practices and interventions available in the community (i.e., the general public have access to it in the community), such as through consultation with a dietician, community care provider, or family physician.
  Arms: Phase 2: Control group Arm

SUMMARY:
This two-phase, double-blind, balanced, parallel-group randomized controlled trial evaluates the feasibility, usability, engagement, and clinical impact of an app-based adaptation of the Mindfulness-Based Eating Awareness Training (MB-EAT) program for adolescents living with obesity.

MB-EAT, has been shown to reduce binge eating episodes, improve food-related self-control, and decrease depressive symptoms in adults with obesity. The app based program promotes mindful awareness and self-regulation in response to hunger and satiety cues, without caloric restriction.

Youth aged 12-17.5 years who are waitlisted or have recently been waitlisted for treatment at the Centre for Healthy Active Living (CHAL) at the Children's Hospital of Eastern Ontario (CHEO) will be enrolled in a 4-week app-based MB-EAT program (Phase 1, n=10) to evaluate feasibility, usability, and engagement.

Phase 2 is a 12-week randomized controlled trial with 160 participants who will be randomized to the experimental arm (app-based MB-EAT program; 60-90 minutes/week) or an active comparator arm (app-based psychoeducation) to evaluate whether the MB-EAT program improves disinhibited eating. At the end of the intervention, 20 participants will be randomly selected for interviews to explore their experiences with the app.

Additional secondary outcomes in Phase 2 include depressive symptoms, anxiety symptoms, emotion regulation, dispositional mindfulness, food craving, mindful eating, body image, health-related quality of life, impact of weight on quality of life, internalized weight bias, food impulsivity, and food reinforcement.

DETAILED DESCRIPTION:
Childhood obesity rates in Canada have nearly tripled over the past 30 years, with approximately 25% of youth aged 12 to 17 years classified as overweight or obese according to body mass index standards. Obesity is a chronic disease linked to increased cardiometabolic risk, psychological comorbidities, and reduced quality of life. Traditional behavioural interventions targeting diet and movement behaviours remain standard care but show limited long-term efficacy. This two-phase, double-blind, balanced, parallel-group randomized controlled trial evaluates the feasibility, usability, engagement, and clinical impact of an app-based adaptation of the Mindfulness-Based Eating Awareness Training (MB-EAT) program for adolescents living with obesity.

MB-EAT, developed by Dr. Jean Kristeller, has been shown to reduce binge eating episodes, improve food-related self-control, and decrease depressive symptoms in adults with obesity. The program promotes mindful awareness and self-regulation in response to hunger and satiety cues, without caloric restriction. This study adapts MB-EAT for delivery through the AmDTx-Epiq app (Mobio Interactive, Toronto, ON), developed with input from mindfulness-based intervention therapists, patients, and software engineers. The digital format aims to improve accessibility and scalability for youth awaiting clinical care.

Eligibility criteria include youth aged 12-17.5 years who are waitlisted or have recently been waitlisted for treatment at the Centre for Healthy Active Living (CHAL) at the Children's Hospital of Eastern Ontario (CHEO), have access to a mobile or tablet device with internet, the ability to complete the study in English, and willingness to provide consent/assent. Exclusion criteria include current enrollment in psychotherapy or a weight management program, diagnosis of bulimia nervosa (purging subtype), certain neurodevelopmental conditions (i.e., Fetal Alcohol Syndrome, Down Syndrome, Prader-Willi Syndrome, Fragile X Syndrome, autism spectrum disorder), or concussion/brain injury within the past six months.

Phase 1 enrolls 10 participants to deliver a 4-week app-based MB-EAT program. The primary objective is to evaluate feasibility, usability, and engagement, as indicated by self-reported interest, enrollment rate, adherence, acceptance, working alliance, expectancy and belief credibility, engagement metrics, attrition, and identified barriers and facilitators. Acceptability will be measured with the Client Satisfaction Questionnaire (modified), usability with the System Usability Scale (modified), credibility and expectancy with the Credibility and Expectancy Questionnaire, and working alliance with the Working Alliance Inventory for Guided Internet Interventions. Engagement will be tracked via in-app metrics, with adherence defined as logging in at least 50% of the required time. Enrollment and attrition rates will be monitored, and post-intervention interviews will explore questionnaire responses, barriers to compliance, and facilitators of app use. The secondary objective for Phase 1 is to assess whether the MB-EAT program improves disinhibited eating in this clinical youth sample.

Phase 2 is a 12-week randomized controlled trial with 160 participants who will be randomized to the experimental arm (app-based MB-EAT program; 60-90 minutes/week) or an active comparator arm (app-based psychoeducation on nutrition, physical activity, and weight management from public health and clinical guidelines). Both arms follow 12 weekly modules via the same platform. At the end of the intervention, 20 participants will be randomly selected for interviews to explore their experiences with the app. The primary outcome is to evaluate whether the MB-EAT program improves disinhibited eating, measured by the Three-Factor Eating Questionnaire Revised 18 Version 2. The secondary objectives are to continually assess feasibility, usability, and engagement with the app-based MBI program using the same indicators and measures applied in Phase 1.

Additional secondary outcomes in Phase 2 include depressive symptoms, anxiety symptoms, emotion regulation, dispositional mindfulness, food craving, mindful eating, body image, health-related quality of life, impact of weight on quality of life, internalized weight bias, food impulsivity, and food reinforcement.

ELIGIBILITY:
Inclusion Criteria:

* Have access to a mobile/tablet device with internet access
* Are aged 12-17.5 years
* Are waitlisted or have recently been waitlised for treatment at CHAL at CHEO
* Are willing and capable to sign consent/assent forms
* Have the ability to complete the study in English

Exclusion Criteria:

* Are currently enrolled in psychotherapy or a weight management program
* Have previously been diagnosed with Bulimia Nervosa, purging subtype
* Have previously been diagnosed with a condition that may impair cognition and neurodevelopment, particularly Fetal Alcohol Syndrome, Down Syndrome, Prader-Willi Syndrome, and Fragile X Syndrome
* Have previously been diagnosed with ASD
* Have had a concussion or brain injury in the past 6-months.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Acceptability | 1 month
  Acceptability will be measured with a modified version of the client satisfaction questionnaire (CSQ). The CSQ is a valid, reliable, 8-item questionnaire used to measure client satisfaction with a particular program or service. The questionnaire has been modified to assess participant satisfaction with the app and is measured with a Likert scale 1 to 4. Higher scores indicating greater satisfaction.
Phase 1: Usability | 1 month
  Usability of the app will be measured using a modified version of the System Usability Scale (SUS). The SUS is a valid and reliable 10-item measure that is used to assess the usability of a system or program with a Likert scale 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate better usability.
Phase 1: Working alliance | 1 month
  The quality of the working alliance with the AmDTx app will be assessed with the Working Alliance Inventory for guided Internet Interventions (WAI-I). The WAI-I is a validated and reliable 12-item questionnaire rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). The scale has been modified to measure working alliance with the app based MBI. The responses are averaged into a total scale (range 1-5), and two sub-scores: Task and goal agreement with the program (8 items; range 1-5); Bond with the guides (4 items; range 1-5). Higher scores indicate better alliance.
Phase 1: Engagement | 1 month
  Engagement with the MBI will be tracked via data collected from the AmDTx app. Engagement will be measured by logins, the number of completed resilience, relaxation and/or psychoeducation sessions + total number of self-assessments of psychological wellbeing + total number of "mindful minutes" (a composite of meaningful engagement with the digital therapeutic), and overall time spent using "meaningful" features within the AmDTx app. Engagement is automatically and anonymously captured for the 4 weeks (the length of the intervention). "Meaningful" refers to features that provide potential benefit for the patient, but do not include neutral engagement such as time spent on the product home screen.
Phase 1: Adherence | 1 month
  Adherence will be measured by the number of times the participant used the intervention, defined as logging into the application 50% of the required time.
Phase 1: Enrollment and attrition rates | 1 month
  Enrollment and attrition rates will be kept track of using a tracking log.
Phase 1: Barriers and facilitators | 1 month
  The potential usefulness and benefits of AmDTx app will be explored via interviews with participants at the end of the intervention phase (4-week follow up), obtaining patient perspective with the app and their respective thoughts on therapeutic utility.
Phase 2: Disinhibited eating | 24 weeks
  Disinhibited Eating (susceptibility to overeat compulsively) will be measured by the Three-Factor Eating Questionnaire Revised 18 Version 2 (TFEQ-R18 V2) which is a likert scale from 1 (definitely true) to 4 (definitely false). High scores on a scale reflect a higher level of disinhibited eating.

SECONDARY OUTCOMES:
Phase 1: Disinhibited Eating | 1 month
  Disinhibited Eating (susceptibility to overeat compulsively) will be measured by the Three-Factor Eating Questionnaire Revised 18 Version 2 (TFEQ-R18 V2) which is a likert scale from 1 (definitely true) to 4 (definitely false). High scores on a scale reflect a higher level of disinhibited eating.
Phase 1 & 2: Depressive symptoms | 4 weeks & 24 weeks
  Measured with the 10-item Center for Epidemiologic Studies Depression (CES-D-10) questionnaire which is a likert scale from 1 (Rarely or non of the time) to 4 (all of the time). A higher score indicates more severe depressive symptoms.
Phase 1 & 2: Anxiety symptoms | 4 weeks & 24 weeks
  Will be measured with the Generalized Anxiety Disorder-7 (GAD-7) scale which is a likert scale from 0 (not at all) to 3 (nearly every day). A higher score indicates more severe anxiety symptoms.
Phase 1 & 2: Emotional regulation | 4 weeks & 24 weeks
  Will be measured using the Difficulties in Emotion Regulation Scale Short Form (DERS-SF) which is a likert scale from 1 (almost never) to 5 (almost always). Higher scores on the DERS-SF indicate greater difficulties in regulating emotions.
Phase 1 & 2: Dispositional mindfulness | 4 weeks & 24 weeks
  Will be measured with the 14-item Mindful Attention Awareness Scale for Adolescents (MAAS-A) which is a likert scale from 1 (almost always) to 6 (almost never). Higher scores are an indication of higher trait mindfulness.
Phase 1 & 2: Disordered eating | 4 weeks & 24 weeks
  Disordered Eating will be measured by the Three-Factor Eating Questionnaire Revised 18 Version 2 (TFEQ-R18 V2) which is a likert scale from 1 (definitely true) to 4 (definitely false). Higher scores representing greater disordered eating.
Phase 1 & 2: Food craving | 4 weeks & 24 weeks
  Will be measured with the Food Cravings Questionnaire Trait Reduced (FCQ-TR) which is a likert scale from 1 (never) to 6 (always). Higher scores indicating more frequent and intense food cravings.
Phase 1 & 2: Mindful eating | 4 weeks & 24 weeks
  Will be measured with the Mindful Eating Questionnaire for Children (MEQ-C) which is a likert scale 1 (never) to 4 (always). Higher scores on the "Mindless Eating" subscale indicate less mindful eating, while higher scores on the "Awareness" subscale indicate more mindful eating.
Phase 1 & 2: Body image | 4 weeks & 24 weeks
  Will be evaluated using the Body Esteem Scale for Adults and Adolescents (BESAA) which is a likert scale 1 (never) to 5 (always). Higher scores indicate higher body esteem.
Phase 2: Enrollment and attrition rates | 12 weeks
  Enrollment and attrition rates will be kept track of using a tracking log.
Phase 2: Adherence | 12 weeks
  Adherence will be measured by the number of times the participant used the intervention, defined as logging into the application 50% of the required time.
Phase 2: Engagement | 12 weeks
  Engagement with the MBI will be tracked via data collected from the AmDTx app. Engagement will be measured by logins, the number of completed resilience, relaxation and/or psychoeducation sessions + total number of self-assessments of psychological wellbeing + total number of "mindful minutes" (a composite of meaningful engagement with the digital therapeutic), and overall time spent using "meaningful" features within the AmDTx app. Engagement is automatically and anonymously captured for the 12 weeks (the length of the intervention). "Meaningful" refers to features that provide potential benefit for the patient, but do not include neutral engagement such as time spent on the product home screen.
Phase 2: Working alliance | 12 weeks
  The quality of the working alliance with the AmDTx app will be assessed with the Working Alliance Inventory for guided Internet Interventions (WAI-I). The WAI-I is a validated and reliable 12-item questionnaire rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). The scale has been modified to measure working alliance with the app based MBI. The responses are averaged into a total scale (range 1-5), and two sub-scores: Task and goal agreement with the program (8 items; range 1-5); Bond with the guides (4 items; range 1-5). Higher scores indicate better alliance.
Phase 2: Barriers and facilitators | 12 weeks
  The potential usefulness and benefits of AmDTx app will be explored via interviews with participants at the end of the intervention phase (12-week follow up), obtaining patient perspective with the app and their respective thoughts on therapeutic utility.
Phase 2: Usability | 12 weeks
  Usability of the app will be measured using a modified version of the System Usability Scale (SUS). The SUS is a valid and reliable 10-item measure that is used to assess the usability of a system or program with a Likert scale 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate better usability.
Phase 2: Acceptability | 12 weeks
  Acceptability will be measured with a modified version of the Client Satisfaction Questionnaire (CSQ). The CSQ is a valid, reliable, 8-item questionnaire used to measure client satisfaction with a particular program or service. The questionnaire has been modified to assess participant satisfaction with the app and is measured with a Likert scale 1 to 4. Higher scores indicating greater satisfaction.
Phase 1 & 2: Health-related quality of life | 4 weeks & 24 weeks
  Will be assessed by the Pediatric Quality of Life (PEDSQL-Adolescent version) which is a likert scale 0 (never) to 4 (almost always). Higher scores indicating better quality of life.
Phase 1 & 2: Impact of weight on quality of life | 4 weeks & 24 weeks
  Will be assessed by the Impact of Weight on Quality of Life - Kids version (IWQOL-Kids) questionnaire which is a likert scale 1 (always true) to 5 (never true). Higher scores indicating a better weight-related quality of life.
Phase 1 & 2: Internalized weight bias | 4 weeks & 24 weeks
  Will be assessed using the Weight Bias Internalization Scale for Youth which is a likert scale 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate a higher level of weight bias internalization.
Phase 1 & 2: Energy intake | 4 weeks & 24 weeks
  As assessed objectively by ad-libitum and by a 3-day self-report journal.
Phase 1 & 2: Food impulsivity | 4 weeks & 24 weeks
  Will be measured with a food-specific impulsivity paradigm based on the Affective Shifting Task (AST).
Phase 1 & 2: Food reinforcement | 4 weeks & 24 weeks
  Measured by a progressive ratio computer task.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Goldfield, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada